CLINICAL TRIAL: NCT02190708
Title: A Phase I, Open Label Study to Assess the Effects of PQ912 on the Pharmacokinetics of Midazolam and Omeprazole in Healthy Male Subjects
Brief Title: Effects of PQ912 on the Pharmacokinetics of Midazolam and Omeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vivoryon Therapeutics N.V. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1002308-8302860; 2014-001883-36 (EudraCT Number)
Record Dates: First submitted 2014-07-04; First posted 2014-07-15 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers; Pharmacologic Action
Keywords: PQ912; Midazolam; Omeprazole; Pharmacokinetics; Drug Interaction
MeSH Terms: interventions — Midazolam; Benzodiazepines; Omeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PQ912 & Midazolam & Omeprazole (Experimental): day2 - day6 800mg PQ912 twice per day po day1 / day6 2.5 mg Midazolam once per day day1 / day6 20 mg Omeprazole once per day
  Interventions: Drug: PQ912; Drug: Midazolam; Drug: Omeprazole

INTERVENTIONS:
Drug: PQ912 — from day2 up to day6 twice daily oral dose of PQ912
  Other Names: Glutaminyl Cyclase Inhibitor
Drug: Midazolam — single oral dose on day1 and day 6
  Other Names: benzodiazepine
Drug: Omeprazole — single oral dose on day1 and day6
  Other Names: Proton pump inhibitor

SUMMARY:
Midazolam is a rapid-acting benzodiazepine, with a short half-life (approximately 1.9 hours) and is primarily metabolised by CYP3A.

Omeprazole is a selective proton pump inhibitor substrate used to reduce gastric acid secretion. Omeprazole is primarily metabolised by CYP2C19.

Midazolam and omeprazole are both used as probe drugs in clinical pharmacology studies to evaluate clinical CYP3A and CYP2C19 drug interactions, respectively. Furthermore the EMA and the FDA guidance on drug interactions recommend the use of these drugs for such evaluations.

The aim of this study is to assess the effect of PQ912 on the PK of midazolam and omeprazole. In vitro studies have demonstrated that PQ912 inhibits several CYP enzymes, including CYP3A4 and CYP2C19 and at the expected exposure levels in patients, has the potential to inhibit these enzymes in-vivo. This study is therefore planned to investigate the potential changes in the PK of midazolam and omeprazole due to the effect of PQ912 at steady-state. In clinical practice it is likely that co-administration of PQ912 with other drugs that are metabolised via the CYP3A and/or CYP2C19 enzymes will occur. This study will provide important information for the requirement of dose adjustments or contraindications in these circumstances.

DETAILED DESCRIPTION:
This will be an open-label, crossover, fixed sequence study in healthy male subjects. Thirty six (36) subjects will participate in the study and will be enrolled as two groups of 18 (Groups 1 and 2).

If the PK data from Group 1 demonstrate a clinically important inhibition of the CYP3A4 and/or CYP2C19 enzymes then the second optional group (Group 2) might be studied at a lower dose level of PQ912 .

Each subject will participate in one treatment period, residing at the CRU from Day -1 (the day before dosing) to Day 7 (until after the last PK sampling occasion).

All subjects will return for a post study visit 5 to 7 days after their final dose.

Dose Regimen:

Each subject will receive single oral doses of midazolam and omeprazole on the morning of Day 1.

On the morning of Day 2, all subjects will commence the multiple dose regimen for PQ912, which will continue for 5 days in total.

Subjects in Group 1 and (if it necessary) in Group 2 will receive PQ912 twice daily (bid) on Days 2 to 6 inclusive and subjects in Group 2 will receive PQ912 bid on Days 2 to 6 inclusive.

On the morning of Day 6 subjects will be given single oral doses of midazolam and omeprazole co-administered with PQ912.

ELIGIBILITY:
Inclusion Criteria:

* males
* of any ethnic origin
* between 18 and 55 years of age
* body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive
* body weight between 50 kg and 100 kg inclusive
* must be in good health,
* will have given written informed consent and to abide by the study restrictions

Exclusion Criteria:

* history of any clinically significant disease or disorder which, in the opinion of the Investigator, may put the subject at risk because of participation in the study, may influence the results, or may limit the subject's ability to participate in the study
* history or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* active participation in a clinical study or participation in a clinical study investigating a new chemical entity within 3 months or 5 half-lives (whichever is longer prior to first dose)
* clinically significant illness within 4 weeks of the start of the dose administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Effect of PQ912 at steady state on pharmacokinetic profile of Omeprazole and Midazolam | from day 1 up to day 6
  Serial blood samples on day 1 and day 6 from predose up to 24 hours postdose

SECONDARY OUTCOMES:
Safety and tolerability of PQ912 in terms of Adverse Events Assessments when coadministered with Midazolam and Omeprazol | day-1 up to day 6 and post dose visit
  Safety profile in terms of Adverse Events Assessments
Safety and tolerability in terms of vital signs (blood pressure, pulse rate, respiration rate, Body temperature) | from baseline up to end of study visit (2 weeks after first treatment)
Safety and Tolerability by assessing changes in electrocardiogram (ECG) parameters | from baseline up to end of study visit (2 weeks after first treatment)
Safety and tolerability in terms of lab tests assessment (hematology, Serum biochemistry, serology, urinalysis) | from baseline up to end of study visit (2 weeks after first treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chiesa, MD, Dr, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom